CLINICAL TRIAL: NCT06370676
Title: Accuracy of Core Body Temperature Measurement Depending on Oesophageal Probe Tip Location
Acronym: ESO-TIP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Mountain Emergency Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: ESO-TIP
Record Dates: First submitted 2024-04-11; First posted 2024-04-17 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Emergencies; Hypothermia
MeSH Terms: conditions — Emergencies; Hypothermia

STUDY DESIGN:
Who Masked: Participant
Masking Description: The participant is blinded for the location of the oesophageal temperature probe tip.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Correctly placed oesophageal probe at +20 degrees celsius ambient temperature (Active Comparator): Oesophageal probe tip located in the lower third of the oesophagus, i.e. behind the left atrium, +20°C ambient temperature, outside terraXcube
  Interventions: Diagnostic Test: Oesophageal temperature measurement
- Oesophageal probe tip too high at +20 degrees celsius ambient temperature (Experimental): Oesophageal probe tip located too high the oesophagus, i.e. behind the trachea, 1-2 cm above the level of the tracheal bifurcation, +20°C ambient temperature, outside terraXcube
  Interventions: Diagnostic Test: Oesophageal temperature measurement
- Correctly placed oesophageal probe at -20 degrees celsius ambient temperature (Active Comparator): Oesophageal probe tip located in the lower third of the oesophagus, i.e. behind the left atrium, -20°C ambient temperature, inside terraXcube
  Interventions: Diagnostic Test: Oesophageal temperature measurement
- Oesophageal probe tip too high at -20 degrees celsius ambient temperature (Experimental): Oesophageal probe tip located too high the oesophagus, i.e. behind the trachea, 1-2 cm above the level of the tracheal bifurcation, -20°C ambient temperature, inside terraXcube
  Interventions: Diagnostic Test: Oesophageal temperature measurement

INTERVENTIONS:
Diagnostic Test: Oesophageal temperature measurement — Oesophageal temperature measurement

SUMMARY:
Background An accurate measurement of the core body temperature (CBT) is of pivotal importance in the management of severely hypothermic patients. For instance, triage decisions for or against extracorporeal rewarming of hypothermic patients in cardiac arrest strongly depend on CBT. CBT measurement with an oesophageal probe is currently considered the gold standard in hypothermic patients with a secured airway in the prehospital setting, with the tip of the probe placed into the distal third of the oesophagus (i.e., posteriorly to the heart and distal to the tracheal bifurcation). However, the correct placement of the probe tip cannot be verified in the prehospital setting, and it is unknown how incorrect placement affects temperature readings.

Hypothesis and aim The investigators hypothesise that an incorrect placement of the oesophageal temperature probe tip could lead to inaccurate measurements (i.e., temperature readings not reflecting the real CBT). Particularly, a tip location too high in the oesophagus in close proximity to the trachea could lead to falsely low temperature readings, especially when the patient is ventilated with cold air. The aim of the proposed study is to investigate the influence of oesophageal temperature probe tip location on CBT measurement.

Methods Experimental, interventional study on 16 healthy volunteers. During the test oesophageal temperature is measured while participants are breathing ambient air first at 20°C (baseline) followed by cold (-20°C) ambient air in supine position for 20 minutes each test in an environmental simulator (terraXcube). Each participant repeats the 20-min test two times with the oesophageal temperature probe tip placed either in the lower third of the oesophagus (i.e., correct position) or too high in the oesophagus, i.e. behind the trachea.

ELIGIBILITY:
Inclusion Criteria:

* Volunteers with an American Society of Anaesthesiologists (ASA) score ≤2.

Exclusion Criteria:

* ASA >3
* Age < 18 and age >75
* Pregnant women
* No signed informed consent
* Signs and symptoms of an acute illness on the study day
* History of oesophageal and nasopharyngeal disorders
* Allergies to Local Anaesthetics (i.e. Lidocain).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2024-05-23 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Difference in core body temperature between the two tip positions | 20 minutes after cold air exposure
  Difference in core body temperature between the two tip positions (i.e. in the lower third of the oesophagus (behind the left atrium) and in the middle third of the oesophagus (behind the trachea)

CONTACTS AND LOCATIONS:
Overall Officials: Simon Rauch, MD, PhD, Principal Investigator — Institute of Mountain Emergency Medicine, Eurac Research
Locations (1):
- TerraXCube, Bolzano, Italy

IPD SHARING:
Plan to Share IPD: No